CLINICAL TRIAL: NCT00004500
Title: A Multicenter, Randomized, Controlled Trial Comparing the Safety and Effectiveness of Bronchoalveolar Lavage With Lucinactant to Standard Care for the Treatment of the Meconium Aspriation Syndrome (MAS) in Newborn Infants
Brief Title: Phase III Randomized Study of Lucinactant in Full Term Newborn Infants With Meconium Aspiration Syndrome
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Slow enrollment and administrative reasons
Sponsor: Windtree Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KL4-MAS-03; FD-R-001938 (Other Grant/Funding Number: US Department of Health and Human Services)
Record Dates: First submitted 1999-10-18; First posted 1999-10-19 (Estimated); Results first posted 2012-05-01 (Estimated); Last update posted 2012-05-03 (Estimated); Status verified 2012-05

CONDITIONS: Meconium Aspiration
Keywords: cardiovascular and respiratory diseases; meconium aspiration syndrome; rare disease
MeSH Terms: conditions — Meconium Aspiration Syndrome; Respiratory Tract Diseases; Rare Diseases | interventions — lucinactant; Surface-Active Agents; Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Lucinactant (Experimental): Lucinactant via bronchoaveolar lavage
  Interventions: Drug: Lucinactant
- Standard Care (Other): Standard Care included the use of oxygen, CMV, sedation, paralysis, vasopressors, and/or alkalinization
  Interventions: Other: Standard Care

INTERVENTIONS:
Drug: Lucinactant — Lucinactant suspension was administered as 10 mg total phospholipid (TPL)/mL, by bronchoalveolar lavage within 90 minutes of randomization. The dose was determined based on the infant's body weight such that the total dose was 16 mL/kg for each of the 2 lavage procedures and 32 mL/kg overall. Infants received 2 doses of lucinactant. Each dose consisted of separate lavage procedures for each lung within 15 minutes (up to 60 minutes) of each other.
  Other Names: Surfactant; KL₄Surfactant
  Arms: Lucinactant
Other: Standard Care — The Standard Care (SC) group received therapies including, but not limited to, the use of oxygen, controlled mechanical ventilation (CMV), sedation, paralysis, vasopressors, and/or alkalinization. The use of adjunctive therapies (namely: high frequency oscillatory ventilation, high frequency jet ventilation, bolus surfactant, inhaled nitric oxide, extra-corporeal membrane oxygenation, or systemic corticosteroids) were not included in SC
  Other Names: Negative Control
  Arms: Standard Care

SUMMARY:
OBJECTIVES:

Evaluate the safety and efficacy of lucinactant administered by bronchoalveolar lavage (BAL) in the treatment of meconium aspiration syndrome (MAS) in newborn infants.

DETAILED DESCRIPTION:
PROTOCOL OUTLINE:

This is a randomized, multicenter study. Patients are randomized to one of two treatment arms.

Arm I: Patients receive lucinactant by bronchoalveolar lavage, into the right and left lung, followed by lung drainage. Treatment repeats when patient stabilizes or every 15 minutes for 2 courses.

Arm II: Patients receive standard treatment including oxygen, conventional mechanical ventilation, sedation, paralysis, vasopressors, and alkalinization.

Patients are followed for 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of meconium aspiration syndrome (MAS)
* Continuous mechanical ventilation (CMV) at time of entry
* Enrollment within 48 hours of birth
* Gestational age of ≥ 37 weeks
* Oxygenation index of ≥ 5 and ≤ 30
* Written informed consent signed and dated by the infant's parent(s) or legal guardian(s)

Exclusion Criteria:

* Congenital anomalies likely to affect any primary or secondary endpoints
* Uncontrollable air leaks
* Hydrops fetalis
* Rupture ≥ 3 weeks of the fetal membranes
* Evidence of overwhelming bacterial infection at time of randomization
* Markedly labile persistent pulmonary hypertension at time of randomization
* Profound neurologic manifestations
* Sustained postductal SpO₂of < 87% for ≥ 15 minutes at an FiO₂of 1.00

Max Age: 48 Hours | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 69 (Actual)
Dates: Start 2000-03; Primary Completion 2002-11 (Actual); Study Completion 2004-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Thomas E Wiswell, Study Chair — Windtree Therapeutics
Locations (1):
- Discovery Laboratories, Inc., Warrington, Pennsylvania, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment occurred between March 2000 and October 2002. Infants were enrolled from neonatal intensive care units and were randomized to open-label study treatment.
Period: Overall Study
Arm/Group | Lucinactant | Standard Care
Started | 38 | 31
1 Year Follow-Up | 24 | 24
Completed | 38 | 31
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Lucinactant | Standard Care | Total
Number analyzed (Participants) | 38 | 31 | 69
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 38 | 31 | 69
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 15 | 31
  Male | 22 | 16 | 38
Region of Enrollment [Number; unit: participants]
  United States | 38 | 31 | 69
Gestational Age [Mean (Standard Deviation); unit: weeks] | 40.0 (1.30) | 39.7 (1.09) | 39.9 (1.21)

OUTCOME MEASURES:

1. Primary Outcome: Number of Days Receiving Mechanical Ventilation (MV)
Description: A patient is not receiving MV if he/she is removed from the mechanical ventilator for ≥ 24 hours. If a patient subsequently requires intubation and MV, the additional time will count as days receiving MV.
Time Frame: 28 days
Population: Data from the initial Phase 1/2 trial were used to estimate the number of subjects required for testing the null hypothesis of no difference between treatment groups. A sample size of 100 subjects per group is required to test the hypothesis at a significance level of 0.05 with a power of 80%.
  All enrolled infants were analyzed (intent-to-treat).
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Lucinactant | Standard Care
Number analyzed (Participants) | 38 | 31
days | 10.2 (9.96) | 8.1 (8.52)

2. Secondary Outcome: Incidence of Death
Time Frame: 28 days
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Lucinactant | Standard Care
Number analyzed (Participants) | 38 | 31
participants | 0 | 0

3. Secondary Outcome: Number of Participants With Air Leaks
Description: Includes pulmonary interstitial emphysema (PIE), Pneumothorax, Pneumomediastinium, and Pneumopericardium
Time Frame: 28 days
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Lucinactant | Standard Care
Number analyzed (Participants) | 38 | 31
participants | 2 | 0

ADVERSE EVENTS:
Time Frame: 28 Days
Description: AEs followed until resolution or stable condition
Arm/Group | Lucinactant | Standard Care
Serious Adverse Events (participants affected / at risk) | 23/38 | 14/31
Other Adverse Events (participants affected / at risk) | 36/38 | 25/31
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Lucinactant (N=38) | Standard Care (N=31)
Bradycardia NOS (Cardiac disorders) | 1 | 0
Cardiac arrest (Cardiac disorders) | 1 | 0
Cardiac tamponade (Cardiac disorders) | 1 | 1
Cardiomyopathy NOS (Cardiac disorders) | 0 | 1
Dysphagia (Gastrointestinal disorders) | 1 | 0
Drug withdrawal syndrome (General disorders) | 2 | 1
Pyrexia (General disorders) | 1 | 0
Oxygen saturation decreased (Investigations) | 1 | 0
Acid-base balance disorder mixed (Metabolism and nutrition disorders) | 1 | 0
Feeding Disorder NOS (Metabolism and nutrition disorders) | 1 | 0
Food intolerance NOS (Metabolism and nutrition disorders) | 0 | 1
Renal impariment NOS (Renal and urinary disorders) | 2 | 0
Renal infarct (Renal and urinary disorders) | 0 | 1
Bronchopulmonary dysplasia (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 11 | 6
Meconium aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pneumothorax NOS (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary Haemorrhage (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Respiratory failure (exc neonatal) (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Stridor (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Hypertension NOS (Vascular disorders) | 1 | 0
Hypotension NOS (Vascular disorders) | 6 | 7
Intraventricular haemorrhage NOS (Vascular disorders) | 0 | 1
Pulmonary hypertension NOS (Vascular disorders) | 11 | 10
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Lucinactant (N=38) | Standard Care (N=31)
Anemia NOS (Blood and lymphatic system disorders) | 5 | 5
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 2 | 0
Thrombocyptopenia (Blood and lymphatic system disorders) | 6 | 2
Bradycardia NOS (Cardiac disorders) | 2 | 1
Cardiomegaly NOS (Cardiac disorders) | 0 | 2
Pulmonary edema NOS (Cardiac disorders) | 2 | 0
Tachycardia NOS (Cardiac disorders) | 2 | 2
Tricuspid valve incompetence (Cardiac disorders) | 0 | 2
Patent ductus arteriosus (Congenital, familial and genetic disorders) | 1 | 3
Drug withdrawn syndrome (General disorders) | 4 | 2
Oedema NOS (General disorders) | 3 | 2
Pyrexia (General disorders) | 2 | 1
Jaundice NOS (Hepatobiliary disorders) | 1 | 2
Pneumonia NOS (Infections and infestations) | 2 | 0
Sepsis NOS (Infections and infestations) | 9 | 3
Blood magnesium decreased (Investigations) | 4 | 1
Oxygen saturation decreased (Investigations) | 4 | 1
Feeding disorder NOS (Metabolism and nutrition disorders) | 6 | 1
Hypocalcemia (Metabolism and nutrition disorders) | 7 | 1
Hypoglycemia NOS (Metabolism and nutrition disorders) | 2 | 0
Hypokalemia (Metabolism and nutrition disorders) | 4 | 5
Hyponatremia (Metabolism and nutrition disorders) | 4 | 4
Hypertonia (Nervous system disorders) | 2 | 0
Hypotonia (Nervous system disorders) | 3 | 0
Oliguria (Renal and urinary disorders) | 4 | 2
Renal impairment NOS (Renal and urinary disorders) | 3 | 0
Atlectasis (Respiratory, thoracic and mediastinal disorders) | 5 | 4
Bronchopulmonary dysplasia (Respiratory, thoracic and mediastinal disorders) | 3 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 19 | 11
Pneumothorax NOS (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 4 | 1
Respiratory failure (exc neonatal) (Respiratory, thoracic and mediastinal disorders) | 3 | 4
Stridor (Respiratory, thoracic and mediastinal disorders) | 2 | 3
Tachypnea (Respiratory, thoracic and mediastinal disorders) | 2 | 3
Rash erythematous (Skin and subcutaneous tissue disorders) | 0 | 2
Procedural site reaction (Surgical and medical procedures) | 2 | 2
Hypertension NOS (Vascular disorders) | 7 | 1
Hypotension NOS (Vascular disorders) | 20 | 13
Pulmonary hypertension NOS (Vascular disorders) | 15 | 11

LIMITATIONS AND CAVEATS:
Early termination led to a small number of subjects analyzed. Results should be interpreted with caution.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days